CLINICAL TRIAL: NCT01272973
Title: Investigation on Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Doses of a Long-acting GLP-1 Analogue in Healthy Male Subjects
Brief Title: Investigation on Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NN9924 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9924-3692; U1111-1118-0257 (Other: Who); 2010-019951-23 (EudraCT Number)
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Oral 1 (Experimental)
  Interventions: Drug: semaglutide; Drug: placebo
- Oral 2 (Experimental)
  Interventions: Drug: semaglutide; Drug: placebo
- Oral 3 (Experimental)
  Interventions: Drug: semaglutide; Drug: placebo
- S.c. (Active Comparator)
  Interventions: Drug: semaglutide

INTERVENTIONS:
Drug: semaglutide — Semaglutide (oral) administered once daily for 10 weeks.Individually adjusted dose investigated up to maximum level.
  Arms: Oral 1; Oral 2; Oral 3
Drug: placebo — Placebo (oral) administered once daily for 10 weeks.
  Arms: Oral 1; Oral 2; Oral 3
Drug: semaglutide — Administered s.c. (under the skin) once weekly for 10 weeks. Individually adjusted dose investigated up to maximum level.
  Other Names: NN9924
  Arms: S.c.

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate safety, tolerability, pharmacokinetics (the rate at which the body eliminates the trial drug) and pharmacodynamics (the effect of the investigated drug on the body) of NN9924 in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, based on an assessment of medical history, physical examination and
* BMI between 21 and 30 kg/m2 (21 inclusive)

Exclusion Criteria:

* Male subjects who are sexually active and unwilling to use a highly effective method of contraception for both them and their nonpregnant partner
* Any clinically significant, abnormal disease history of the following systems: cardio-pulmonary, gastrointestinal, hepatic, neurological, renal,genitourinary, endocrine or haematological
* The receipt of any investigational product within 90 days before screening, or is currently enrolled in any other clinical trial

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) | from the first trial related activity (screening visit) and until completion of the post treatment follow-up visit 91-105 days after first dose

SECONDARY OUTCOMES:
Hypoglycaemic episodes | from the first trial related activity (screening visit) and until completion of the post treatment follow-up visit 91-105 days after first dose
Laboratory safety variables (haematology, biochemistry, and urinalysis) | from the first trial related activity (screening visit) and until completion of the post treatment follow-up visit 91-105 days after first dose
Maximum plasma concentration of NN9924 | after dosing on the 68th, 69th and 70th Day
Area under the plasma concentration curve over the dosing interval (0-24 hours) | after dosing on the 68th, 69th and 70th day
Terminal phase elimination half-life | from last dose (day 70) to follow-up visit 91-105 days after first dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Berlin, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com